CLINICAL TRIAL: NCT01551849
Title: Echocardiographic Assessment of Function During ECMO Support
Status: Completed | Type: Observational
Sponsor: Nationwide Children's Hospital (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor
Other Study IDs: IRB11-00470; 12CRP9020022 (Other Grant/Funding Number: AHA 12CRP9020022)
Record Dates: First submitted 2012-03-09; First posted 2012-03-13 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Cardiac Failure; Extracorporeal Membrane Oxygenation Complication
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- VA-ECMO patients: Patients placed on VA-ECMO support for primary cardiac dysfunction.

SUMMARY:
The purpose of this study is to evaluate echocardiographic markers of cardiac function to assess the ability of patients to successfully end VA-ECMO support.

DETAILED DESCRIPTION:
1. What is the major problem being addressed by this study?

   Extracorporeal membrane oxygenation (ECMO) is a machine used to do the work of the heart and lungs when children's hearts or lungs are too sick to perform normally. Veno-arterial (VA) ECMO therapy for poor heart function provides support that can lead to patient recovery, transplantation if appropriate and eligible, or complications of ECMO therapy lead to stopping care. Each day a patient is on ECMO, complications can occur that require stopping support, and attempting to get off ECMO as quickly as possible is important. There is currently no consistent way of assessing heart function while patients are supported by VA-ECMO to help guide when children's hearts have improved enough to survive without the help of ECMO.
2. What specific questions are you asking and how will you attempt to answer them?

The specific question we are asking is whether newer ultrasound measures of heart function can predict which patient may be well enough to be able to come off of ECMO support. We are following critically ill patients and performing multiple measurements at specific time points to look for changes in those patients whose heart function recovers and in those patients who do not recover function. The ultrasound measurements will be performed during changes in the amount of support provided by the ECMO machine.

* 3. What is the long-term biomedical significance of your work, particularly as it pertains to the cardiovascular area? What major therapeutic advance(s) do you anticipate that it will lead to? For instance, new drug(s), a surgical technique/procedure, a diagnostic tool/test, a previously undetected risk factor, etc.

Our long term goal is to develop non-invasive, quantitative measures of cardiac function for patients needing ECMO support to help guide care. Ultimately if deemed successful, these measurements could be used by all physicians who care for these patients. This study could lead to more efficient prediction of who needs to stay on ECMO and who could be removed. This could help to improve survival and decrease complications in some of the sickest children. These measurements may also help us to identify, at an early stage, those patients whose hearts are too sick to recover and will need a heart transplant evaluation.

ELIGIBILITY:
Inclusion Criteria:

* VA ECMO (all cannulation sites)
* Primary Cardiac Failure
* Septic Shock

Exclusion Criteria:

* VV ECMO
* Primary Respiratory Failure
* Congenital Diaphragmatic Hernia
* Persistent pulmonary hypertension of the newborn
* greater than 1 source of systemic perfusion

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Critically ill patients supported by VA-ECMO in the NICU, PICU, or CTICU.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2016-12-30 (Actual); Study Completion 2016-12-30 (Actual)

PRIMARY OUTCOMES:
Ability to separate from VA-ECMO support with stable hemodynamics | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Andrew R Yates, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
non-interventional trial